CLINICAL TRIAL: NCT06363968
Title: Electroretinogram (ERG) as a Potential Biomarker of Serotonin Selective Reuptake Inhibitor (SSRI)-Responsive Posttraumatic Stress Disorder (PTSD): A Pilot Study
Brief Title: Biomarkers in the Retina for Prognosticating Mental Health Treatments
Acronym: BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1743326
Record Dates: First submitted 2024-03-18; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: PTSD; Posttraumatic Stress Disorder
Keywords: PTSD; posttraumatic stress disorder; SSRI; antidepressant; serotonin; electroretinogram; ERG
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Electroretinography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ERG, all participants (Experimental): All participants undergo ERG recording before and after a single dose of sertraline 50 mg.
  Interventions: Device: RETeval

INTERVENTIONS:
Device: RETeval — as previous
  Other Names: electroretinogram; ERG

SUMMARY:
Title: ERG as a potential biomarker of SSRI-responsive PTSD: A pilot study

Posttraumatic stress disorder (PTSD) affects many individuals who experience a traumatic event. Previous studies suggest that there is a connection between the brain and the retina, and that the electroretinogram (ERG) may be a valuable biomarker to tell us more about signals in the brain that are related to mental health disorders like PTSD. The goal of this observational study is to examine the ERG waveform in veterans with PTSD before and after a single dose of the selective serotonin reuptake inhibitor (SSRI), sertraline. Sertraline is one of two FDA-approved medications for the treatment of PTSD. The main questions this pilot study aims to answer are:

1. How does sertraline, an SSRI, influence the ERG waveform in veterans with PTSD?
2. Is there a significant correlation between baseline ERG signals and the change in ERG following SSRI treatment?

Participants will be asked to:

* Undergo ERG recordings before and after a single dose of sertraline.
* Provide relevant clinical information related to PTSD symptoms and treatment history.

Following the initial study visits, participants will enter an optional open label phase of the study in which qualifying participants who initiate antidepressant treatment through routine clinical care will be invited back for a follow-up ERG recording.

DETAILED DESCRIPTION:
In this study, individuals will undergo an assessment that includes taking a history of their previous exposure to traumatic events, an assessment of current mental health symptoms including those associated with PTSD, and an assessment of physiologic measures, including ERG as well as vital sign measurements, blood draw, and saliva sampling. Participants will be given a single dose of sertraline (50mg), and a repeat ERG will be administered. An optional open label phase of the study will follow, in which participants who undergo treatment with an antidepressant will be invited back for a follow-up assessment with repeat ERG.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the U.S. Armed Forces
* Current diagnosis of PTSD

Exclusion Criteria:

* Known diagnosis of a primary psychotic or major neurocognitive disorder
* Significant bilateral visual loss
* History of acute angle closure glaucoma
* Known inherited retinal disease
* Previous ERG deficits
* Known photosensitive epilepsy
* Known current pregnancy or lactation
* Allergy or previous adverse reaction to sertraline or SSRI
* Allergy to Sensor Strip gel
* Hepatic failure
* Damage to orbit structure or open lesion in soft tissue surrounding the eye
* Any use in the time period of at least 6 half-lives prior to baseline of sertraline or other drugs acting on serotonin and/or unwillingness to avoid these medications for the duration of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
ERG b-wave amplitude response to SSRI | ERGs will be performed at the baseline visit prior to a single dose of sertraline, and again after sertraline the following day. ERG will also be performed at the follow up visit for a subset of participants who qualify, up to 1 year following baseline.
  The change in b-wave amplitude following a single dose of sertraline compared to baseline b-wave amplitude will be calculated. The relationship between baseline b-wave amplitude and change in b-wave amplitude will be analyzed.

SECONDARY OUTCOMES:
Total Clinician Administered PTSD Scale for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition; CAPS-5) score | PTSD measures will be collected as a part of the baseline assessment. CAPS-5 will also be readministered at the follow up visit for a subset of participants who qualify, up to 1 year following baseline.
  CAPS-5 administered at baseline
Total PTSD Checklist for DSM-5 (PCL-5) | PTSD measures will be collected as a part of the baseline assessment. PCL-5 will also be repeated at the follow up visit for a subset of participants who qualify, up to 1 year following baseline.
  Self report PTSD Checklist (PCL-5) administered at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hendrickson, MD, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States